CLINICAL TRIAL: NCT02671968
Title: Real-Time Continuous Glucose Monitoring (RT-CGM) in Patients With Type 1 Diabetes at High Risk for Low Glucose Values Using Multiple Daily Injections (MDI) in Germany (HYPODE-STUDY)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Science Consulting in Diabetes (Industry)
Collaborators: DexCom, Inc. a Delaware corporation, USA (Unknown); Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel
Other Study IDs: IDT-1510-SI / HypoDE
Record Dates: First submitted 2016-01-25; First posted 2016-02-02 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Diabetes
Keywords: CGM; hypoglycemic events
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

ARMS (2):
- CGM group (Experimental)
  Interventions: Device: Continuous Glucose Monitoring System
- Control group (No Intervention)

INTERVENTIONS:
Device: Continuous Glucose Monitoring System
  Other Names: Dexcom G5 Mobile, Dexcom G4
  Arms: CGM group

SUMMARY:
Demonstrate that usage of RT-CGM (Real time continuous glucose monitoring) reduces the frequency of low CGM-recorded glucose events in patients using MDI (Multiple daily injections) that are at risk for hypoglycemic events.

DETAILED DESCRIPTION:
In a randomized controlled trial the primary hypothesis is tested if the usage of RT-CGM in the intervention group (CGM group) reduces the frequency of glucose values <55 mg/dl in patients with hypoglycemia problems (hypoglycemia unawareness or documented previous severe hypoglycemia) significantly more than in the control group receiving usual care (without CGM).

Secondary is tested if patients in the CGM group showed a significantly more favorable change in the below defined secondary endpoint than patients in the control group after 26 weeks follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes for at least 12 months on multiple daily injections (MDI). MDI is defined as prandial insulin injections at each major meal (excludes pre-mixed insulin) with doses determined by SMBG and carbohydrate counting, and basal insulin injection(s)
* Age ≥ 18 years
* HbA1c ≤ 9.0 % performed within 4 months before begin of the study
* High risk for severe hypoglycemia (defined as a score of 4 or higher on the Hypoglycemia unawareness scale (HUS) or a history of at least one severe hypoglycemic event in the last 12 months (required third part assistance, not able to treat themselves))
* Willing to not use paracetamol or drugs containing it
* Signed and dated Informed Consent Form

Exclusion Criteria:

* Use of personal real-time-CGM 3 months prior to study entry and during the study (except study devices)
* Use of a flash-glucose monitoring system 3 months prior to study and during the study
* Alcoholism or drug abuse
* Unable to comply with the protocol at the investigators discretion, such as known psychiatric diagnosis, cognitive / physical decline
* Pregnancy or lactation period
* Severe known allergies, e.g. against plaster
* Mental incapacity or language barriers precluding adequate compliance with the study procedures
* Limited or no legal capacity or legal guardianship
* Dependency from the sponsor or the clinical investigator (e.g. co-workers of the sponsor or the clinical research center or their families)
* Participation in another study at the same time with a non-approved drug or a non-CE-labelled medical device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2016-02; Primary Completion 2017-07-14 (Actual); Study Completion 2017-10-24 (Actual)

PRIMARY OUTCOMES:
Change in the total number of low glucose events (<55 mg/dl), between baseline and outcome phase (week 22-26) in CGM group and control group (change = subtracting number of follow up events from number of baseline events | For each subject, the experimental phase has an expected duration of up to 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Hermanns, Prof., Principal Investigator — Forschungsinstitut Diabetes-Akademie Bad Mergentheim (FIDAM)
Locations (12):
- Germany (12):
  - Gemeinschaftspraxis Dres. Klausmann, Aschaffenburg
  - m&i-Fachklinik Bad Heilbrunn, Bad Heilbrunn
  - Forschungsinstitut Diabetes-Akademie Bad Mergentheim (FIDAM), Bad Mergentheim
  - Diabetologische Schwerpunktpraxis, Bergheim
  - Medicover Berlin-Mitte, Berlin
  - Diabetologikum Duisburg, Duisburg
  - Diabetes Praxis Essen, Essen
  - Diabetologische Schwerpunktpraxis mit Fußambulanz, Essen
  - Zentrum für Diabetologie Bergedorf, Hamburg
  - Gemeinschaftspraxis Dres. Kaltheuner, Leverkusen
  - Diabetes Schwerpunkt Praxis Zentrum für Hormone und Stoffwechsel, Marktredwitz
  - Schwerpunktpraxis für Diabetes und Ernährungsmedizin, Münster

REFERENCES:
- [Derived] Hermanns N, Heinemann L, Kulzer B, Schafer A, Jacobsen M, Ehrmann D. Continuous glucose monitoring as equinox of nocturnal and daytime hypoglycaemia in type 1 diabetes: insights from the randomized controlled HypoDE trial. Diabetes Res Clin Pract. 2025 Jun;224:112228. doi: 10.1016/j.diabres.2025.112228. Epub 2025 May 8. PMID 40348338
- [Derived] Hermanns N, Ehrmann D, Heinemann L, Freckmann G, Waldenmaier D, Calhoun P. Real-Time Continuous Glucose Monitoring Can Predict Severe Hypoglycemia in People with Type 1 Diabetes: Combined Analysis of the HypoDE and DIAMOND Trials. Diabetes Technol Ther. 2022 Sep;24(9):603-610. doi: 10.1089/dia.2022.0130. Epub 2022 Jun 10. PMID 35604794
- [Derived] Waldenmaier D, Freckmann G, Pleus S, Hermanns N, Ehrmann D, Heinemann L, Haug C. Therapy adjustments in people with type 1 diabetes with impaired hypoglycemia awareness on multiple daily injections using real-time continuous glucose monitoring: a mechanistic analysis of the HypoDE study. BMJ Open Diabetes Res Care. 2021 Apr;9(1):e001848. doi: 10.1136/bmjdrc-2020-001848. PMID 33863716
- [Derived] Heinemann L, Freckmann G, Ehrmann D, Faber-Heinemann G, Guerra S, Waldenmaier D, Hermanns N. Real-time continuous glucose monitoring in adults with type 1 diabetes and impaired hypoglycaemia awareness or severe hypoglycaemia treated with multiple daily insulin injections (HypoDE): a multicentre, randomised controlled trial. Lancet. 2018 Apr 7;391(10128):1367-1377. doi: 10.1016/S0140-6736(18)30297-6. Epub 2018 Feb 16. PMID 29459019
- See also: Real-time continuous glucose monitoring in adults with type 1 diabetes and impaired hypoglycaemia awareness or severe hypoglycaemia treated with multiple daily insulin injections (HypoDE): a multicentre, randomised controlled trial. — https://www.ncbi.nlm.nih.gov/pubmed/29459019